CLINICAL TRIAL: NCT02020044
Title: Prospective Clinical Study on Postoperative Outcome After Descemet Membrane Endothelial Keratoplasty (DMEK) and Ultra-thin Descemet Stripping Automated Endothelial Keratoplasty (DSAEK)
Brief Title: Outcome After Descemet Membrane Endothelial Keratoplasty (DMEK) and Ultra-thin Descemet Stripping Automated Endothelial Keratoplasty (DSAEK)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Necip Torun, Necip, Torun, MD, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA2/108/12
Record Dates: First submitted 2013-12-11; First posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Fuchs' Endothelial Corneal Dystrophy; Bullous Keratopathy; Iridocorneal Endothelial Syndrome; Posterior Polymorphous Dystrophy; Endothelial Dysfunction
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Iridocorneal Endothelial Syndrome | interventions — Descemet Stripping Endothelial Keratoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endothelial Keratoplasty (Other): Descemet membrane endothelial keratoplasty DMEK Ultra-thin Descemet stripping automated endothelial keratoplasty Ultra-thin DSAEK
  Interventions: Other: Endothelial Keratoplasty

INTERVENTIONS:
Other: Endothelial Keratoplasty
  Other Names: DMEK; Descemet Membrane Endothelial Keratoplasty; Ultra-thin Descemet stripping automated endothelial keratoplasty; Ultra-thin DSAEK

SUMMARY:
The purpose of this study is evaluate the outcome after posterior lamellar keratoplasty (DMEK and Ultra-thin DSAEK) for corneal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or older
* Scheduled to undergo endothelial keratoplasty
* Able to provide written informed consent.

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity (change from baseline) | 1, 3, 6, and 12 months and annually

SECONDARY OUTCOMES:
Endothelial cell density (change from baseline) | 1, 3, 6, and 12 months and annually
Intraocular pressure (change from baseline) | 1, 3, 6, and 12 months and annually
Manifest refraction (change from baseline) | 1, 3, 6, 12 months and annually
corneal pachymetry (change from baseline) | 1, 3, 6, 12 months and annually
Quality of Life, NEI-VFQ 25 (change from baseline) | 3, 12 months, annualy
  Questionnaire
corneal topography (change from baseline) | 1, 3, 6, and 12 months and annually
Anterior Segment OCT of cornea and anterior chamber angle (change from baseline) | 1, 3, 6, and 12 months and annually
postoperative Medication (change from baseline) | 1,3,6 and 12 months and annually
Histological Sample of Recipient's Descemet Membrane | intraoperative
  Recipient's Descemet Membrane

CONTACTS AND LOCATIONS:
Overall Officials: Necip Torun, MD, Study Director — Department of Ophthalmology, Charité - Unviersitätsmedizin Berlin
Locations (1):
- Department of Ophthalmology, Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Maier AK, Gundlach E, Gonnermann J, Klamann MK, Eulufi C, Bertelmann E, Joussen AM, Torun N. Fellow Eye Comparison of Descemet Membrane Endothelial Keratoplasty and Penetrating Keratoplasty. Cornea. 2013 Oct;32(10):1344-8. doi: 10.1097/ICO.0b013e31829dd816. PMID 23928950
- [Background] Maier AK, Gundlach E, Klamann MK, Gonnermann J, Bertelmann E, Joussen AM, Torun N, Rieck PW. [Influence of donor lamella thickness on visual acuity after Descemet's stripping automated endothelial keratoplasty (DSAEK)]. Ophthalmologe. 2014 Feb;111(2):128-34. doi: 10.1007/s00347-013-2795-0. German. PMID 23575642
- [Background] Maier AK, Klamann MK, Torun N, Gonnermann J, Schroeter J, Joussen AM, Rieck P. Intraocular pressure elevation and post-DSEK glaucoma after Descemet;s stripping endothelial keratoplasty. Graefes Arch Clin Exp Ophthalmol. 2013 Apr;251(4):1191-8. doi: 10.1007/s00417-012-2203-5. Epub 2012 Nov 20. PMID 23180233
- [Background] Guerra FP, Anshu A, Price MO, Giebel AW, Price FW. Descemet's membrane endothelial keratoplasty: prospective study of 1-year visual outcomes, graft survival, and endothelial cell loss. Ophthalmology. 2011 Dec;118(12):2368-73. doi: 10.1016/j.ophtha.2011.06.002. Epub 2011 Aug 27. PMID 21872938
- [Background] van Dijk K, Ham L, Tse WH, Liarakos VS, Quilendrino R, Yeh RY, Melles GR. Near complete visual recovery and refractive stability in modern corneal transplantation: Descemet membrane endothelial keratoplasty (DMEK). Cont Lens Anterior Eye. 2013 Feb;36(1):13-21. doi: 10.1016/j.clae.2012.10.066. Epub 2012 Oct 26. PMID 23108011
- [Derived] Gundlach E, Pilger D, Brockmann T, Dietrich-Ntoukas T, Joussen AM, Torun N, Maier AB. Recovery of Contrast Sensitivity After Descemet Membrane Endothelial Keratoplasty. Cornea. 2021 Sep 1;40(9):1110-1116. doi: 10.1097/ICO.0000000000002686. PMID 33591041
- [Derived] Gundlach E, Spiller N, Pilger D, Dietrich-Ntoukas T, Joussen AM, Torun N, Maier AB. Impact of difficult unfolding and attachment of the graft lamella on the long-term outcome after Descemet membrane endothelial keratoplasty. Graefes Arch Clin Exp Ophthalmol. 2020 Nov;258(11):2459-2465. doi: 10.1007/s00417-020-04852-z. Epub 2020 Jul 23. PMID 32705337
- [Derived] Maier AK, Gundlach E, Pilger D, Rubsam A, Klamann MK, Gonnermann J, Bertelmann E, Joussen AM, Torun N. Rate and Localization of Graft Detachment in Descemet Membrane Endothelial Keratoplasty. Cornea. 2016 Mar;35(3):308-12. doi: 10.1097/ICO.0000000000000740. PMID 26764881
- [Derived] Gonnermann J, Maier AK, Klamann MK, Brockmann T, Bertelmann E, Joussen AM, Torun N. Posterior iris-claw aphakic intraocular lens implantation and Descemet membrane endothelial keratoplasty. Br J Ophthalmol. 2014 Sep;98(9):1291-5. doi: 10.1136/bjophthalmol-2014-304948. Epub 2014 Apr 29. PMID 24782475